CLINICAL TRIAL: NCT06542146
Title: Impact of Dietary Intervention on Children of ADHD at Sohag University Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Bahaa Abdelazeem, assistant lecteurer neuropsychiatry department sohag univerisity hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-07-2MD
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): patients will follow usual diet
  Interventions: Dietary Supplement: Usual diet
- group B (Active Comparator): Patients will follow Mediterranean die
  Interventions: Dietary Supplement: Mediterranean diet

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — The Mediterranean diet is consisting of fruits, vegetables , legumes, whole grains, nuts, and olive oil as the main source ofdietary fat
  Arms: group B
Dietary Supplement: Usual diet — Usual diet including routine diet we already eat
  Arms: group A

SUMMARY:
Attention-deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder of persistent impairment of attention, hyperactivity, and impulsivity which worsens daily functioning and quality of life , including social troubles , poor academic achievement and occupational problems .It is one of the most common psychiatric disorders between children . The prevalence of ADHD was 7.2% all over the world in 2015 and this percentage is increasing every year . In Arab countries, A systematic review of studies reported that the prevalence of ADHD ranged from 1.3% to 16%. . ADHD has been treated with medical treatment such as psychostimulants (methylphenidate and amphetamines), noradrenergic treatment as atomoxetine and alpha-2A-adrenergic agonists as guanfacine and clonidine , behavioral treatment and their combination . Due to adverse effects of medical treatments and behavioral therapy limitations, other approaches to augment multimodal ADHD management has been tested . Non medical treatment as Digital therapeutics may improve cognitive functions and attention in ADHD . Physical activity interventions for ADHD may improve cognitive , physical and psychological functions.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years children with ADHD

Exclusion Criteria:

* patient with eating disorders.

  * patients with chronic medical illness.
  * patients with IQ below 70.
  * patients who would drop out from the study

    1. if patient would be absent for 3 months,
    2. if patient would fail for any reason to continue his dietary restriction.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Severity of ADHD symptoms | 6 months
  WEISS functional impairment rating scale-parent form (WFIRS-P) to assess the severity of ADHD symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polanczyk GV, Willcutt EG, Salum GA, Kieling C, Rohde LA. ADHD prevalence estimates across three decades: an updated systematic review and meta-regression analysis. Int J Epidemiol. 2014 Apr;43(2):434-42. doi: 10.1093/ije/dyt261. Epub 2014 Jan 24. PMID 24464188
- [Background] Christiansen L, Beck MM, Bilenberg N, Wienecke J, Astrup A, Lundbye-Jensen J. Effects of Exercise on Cognitive Performance in Children and Adolescents with ADHD: Potential Mechanisms and Evidence-based Recommendations. J Clin Med. 2019 Jun 12;8(6):841. doi: 10.3390/jcm8060841. PMID 31212854
- [Background] Chen HJ, Lee YJ, Yeh GC, Lin HC. Association of attention-deficit/hyperactivity disorder with diabetes: a population-based study. Pediatr Res. 2013 Apr;73(4 Pt 1):492-6. doi: 10.1038/pr.2013.5. Epub 2013 Jan 17. PMID 23329200
- [Background] Arnold LE, Kleykamp D, Votolato NA, Taylor WA, Kontras SB, Tobin K. Gamma-linolenic acid for attention-deficit hyperactivity disorder: placebo-controlled comparison to D-amphetamine. Biol Psychiatry. 1989 Jan 15;25(2):222-8. doi: 10.1016/0006-3223(89)90167-4. PMID 2539203